CLINICAL TRIAL: NCT00338104
Title: Conversion of Hyperglycemic Patients Being Treated With Intravenous Insulin Infusions to Lantus Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Mark E. Molitch, M.D., Northwestern University Feinberg School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0361-028
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Results first posted 2009-04-06 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-03

CONDITIONS: Hyperglycemia; Diabetes
Keywords: insulin; glargine; intravenous; subcutaneous; hospital; diabetes; glucose; inpatient
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40% Glargine (Experimental): Patients will receive a dose of glargine insulin equal to 40% of insulin drip rate.
  Interventions: Drug: insulin glargine
- 60% Glargine (Experimental): Patients will receive a dose of glargine insulin equal to 60% of insulin drip rate.
  Interventions: Drug: insulin glargine
- 80% Glargine (Experimental): Patients will receive a dose of glargine insulin equal to 80% of insulin drip rate.
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin glargine — Insulin glargine given at 40% of prior stable drip rate.
  Other Names: Lantus is brand name for Glargine
  Arms: 40% Glargine
Drug: insulin glargine — Insulin glargine given at 60% of prior stable drip rate.
  Other Names: Lantus is brand name for Glargine
  Arms: 60% Glargine
Drug: insulin glargine — Insulin glargine given at 80% of prior stable drip rate.
  Other Names: Lantus is brand name for Glargine
  Arms: 80% Glargine

SUMMARY:
The primary objective of this study is to determine the optimal dose of glargine insulin when converting from intravenous short-acting continuous insulin infusions in surgical and intensive care unit patients using a prospective, controlled, parallel group, randomized study design.

Note: Lantus insulin is the proprietary name for glargine insulin.

DETAILED DESCRIPTION:
Critical illness causes an impairment of insulin secretion and insulin action, resulting in hyperglycemia even in normal individuals and a worsening of the hyperglycemia in patients with diabetes. Normalization of elevated glucose levels by intensive insulin infusion therapy in these critically ill patients has been proven to dramatically improve in-hospital mortality rates. After glucose levels have been controlled with insulin infusions, the best way to convert them to subcutaneous insulin regimens has not been demonstrated conclusively but the insulin regimen best suited is a combination of a basal insulin such as glargine (Lantus) insulin with premeal insulin boluses using a short-acting insulin such as Lispro or Aspart.

Subjects will be randomized into three groups, 25 subjects in each group, the groups differing according to the starting dose of glargine insulin as follows:

1. Multiply the total daily IV insulin dose, using the final 6 hour infusion rate to estimate the total daily dose, by 0.4 to get the starting dose of glargine, continuing the insulin drip for 5 hours after giving the glargine before stopping the infusion;
2. Multiply the total daily IV insulin dose, using the final 6 hour infusion rate to estimate the total daily dose, by 0.6 to get the starting dose of glargine, continuing the insulin drip for 5 hours after giving the glargine before stopping the infusion;
3. Multiply the total daily IV insulin dose, using the final 6 hour infusion rate to estimate the total daily dose, by 0.8 to get the starting dose of glargine, continuing the insulin drip for 5 hours after giving the glargine before stopping the infusion.

The glargine insulin will then be continued as the basal insulin, adjusting doses every 24 hours based on the fasting blood glucose level. In addition, patients will receive Lispro or Aspart insulin as prandial bolus insulins with the goals premeal being 80 - 120 mg/dl, including bedtime. Glucose measurements will be obtained every 1- 4 hours while patients are on their insulin infusions, depending upon the stability of their condition and the stability of their glucose levels. Following transfer to glargine insulin, they will have glucose measured at least four times per day, premeal and bedtime as per standard protocol in the hospital for patients receiving insulin. Glucose data will be obtained from such patients and this will be compared among the various glargine regimens.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose > 100 mg/dl
* Patients on surgical services or in intensive care units receiving intravenous insulin

Exclusion Criteria:

* Inability to obtain informed consent from patient or next-of-kin
* Allergy to insulin
* Participation in another research study
* Patients for whom there are "do-not-resuscitate" orders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Molitch, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Schmeltz LR, DeSantis AJ, Schmidt K, O'Shea-Mahler E, Rhee C, Brandt S, Peterson S, Molitch ME. Conversion of intravenous insulin infusions to subcutaneously administered insulin glargine in patients with hyperglycemia. Endocr Pract. 2006 Nov-Dec;12(6):641-50. doi: 10.4158/EP.12.6.641. PMID 17229660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 patients with hyperglycemia were recruited from the inpatient service at Northwestern Memorial Hospital between August, 2004 and May, 2005.
Pre-assignment Details: Patients had to be on a continuous insulin infusion to treat hyperglycemia prior to randomization
Groups:
- 40% Group: Glargine at 40% of insulin drip rate
- 60% Group: Glargine at 60% of insulin drip rate
- 80% Group: Glargine at 80% of insulin drip rate
Period: Overall Study
Arm/Group | 40% Group | 60% Group | 80% Group
Started | 25 | 25 | 25
Completed | 23 | 24 | 22
Not Completed | 2 | 1 | 3
Not completed — Protocol Violation | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40% Group | 60% Group | 80% Group | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (13.7) | 60.7 (10.8) | 58.6 (10.2) | 60.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 7 | 19
  Male | 20 | 18 | 18 | 56
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.9 (5.0) | 30.6 (6.4) | 29.9 (8.0) | 29.8 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Blood Glucose Values Between 80 - 140
Description: Percentage of blood glucose values within the target range of eighty to one hundred forty mg per dL
Time Frame: First 24 hours after conversion
Measure: Number; unit: percentage of blood glucose values
Arm/Group | 40% Group | 60% Group | 80% Group
Number analyzed (Participants) | 23 | 24 | 22
percentage of blood glucose values | 43 | 35 | 48

2. Secondary Outcome: Percentage of Glucose Values < 50 mg/dL
Description: Percentage of blood glucose values < 50 mg/dL
Time Frame: First 24 hours after conversion
Measure: Number; unit: percentage of blood glucose values
Arm/Group | 40% Group | 60% Group | 80% Group
Number analyzed (Participants) | 23 | 24 | 22
percentage of blood glucose values | 1 | 0 | 0

3. Secondary Outcome: Percentage of Glucose Levels > 180 mg/dL
Description: Percentage of blood glucose levels > 180 mg/dL
Time Frame: First 24 hours after conversion
Measure: Number; unit: percentage of blood glucose values
Arm/Group | 40% Group | 60% Group | 80% Group
Number analyzed (Participants) | 23 | 24 | 22
percentage of blood glucose values | 19 | 34 | 18

LIMITATIONS AND CAVEATS:
not all patients were analyzed in each group because insulin not given appropriately to those patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No